CLINICAL TRIAL: NCT02301039
Title: SARC028: A Phase II Study of the Anti-PD1 Antibody Pembrolizumab (MK-3475) in Patients With Advanced Sarcomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sarcoma Alliance for Research through Collaboration (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SARC028
Record Dates: First submitted 2014-11-17; First posted 2014-11-25 (Estimated); Results first posted 2020-09-29 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Soft Tissue Sarcoma; Bone Sarcoma
MeSH Terms: conditions — Sarcoma; Bone Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Soft tissue sarcoma (Experimental): Patients with the following types of soft tissue sarcoma: leiomyosarcoma, poorly differentiated/de-differentiated liposarcoma, high grade pleomorphic undifferentiated sarcoma/MFH, MPNST and synovial sarcoma). Pembrolizumab will be administered at 200 mg intravenously every 3 weeks
  Interventions: Drug: Pembrolizumab
- Bone sarcoma (Experimental): Patients with the following types of bone sarcoma: Ewing sarcoma, osteosarcoma, and chondrosarcoma [de-differentiated or mesenchymal]. Pembrolizumab will be administered at 200 mg intravenously every 3 weeks
  Interventions: Drug: Pembrolizumab
- Expansion (Experimental): Patients with the following types of soft tissue sarcoma: poorly differentiated/de-differentiated liposarcoma, high grade pleomorphic undifferentiated sarcoma. Pembrolizumab was administered at 200 mg intravenously every 3 weeks
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab
  Other Names: Mk-3475

SUMMARY:
The purpose of this study is to determine the efficacy of pembrolizumab in patients with advanced sarcomas.

DETAILED DESCRIPTION:
This is a multi-institutional phase II study of pembrolizumab in patients with advanced sarcomas. This study will have two treatment groups, one group for patients with soft tissue sarcoma and one group for patients with bone sarcoma.

Initial enrollment for this study included a total of 86 patients with soft tissue sarcoma and bone sarcomas.

In the expansion portion, there will be an additional 30 patients with undifferentiated pleomorphic sarcoma (UPS) and 30 patients with dedifferentiated or other high grade liposarcoma (LPS) enrolled into the study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years (Age ≥ 12 years for patients with bone sarcomas).
* Histologically confirmed diagnosis of unresectable, recurrent, and/or metastatic high grade soft-tissue or bone sarcoma of one of the following subtypes: soft tissue sarcomas (leiomyosarcoma, poorly differentiated/de-differentiated liposarcoma, high grade pleomorphic undifferentiated sarcoma/MFH and synovial sarcoma), and bone sarcomas (Ewing sarcoma, osteosarcoma, and chondrosarcoma [de-differentiated or mesenchymal]).
* ECOG Performance Status of 0 or 1.
* At least one site of measurable disease on CT/MRI scans as defined by RECIST 1.1. Baseline imaging must be performed within 30 days of dosing.
* At least one site of accessible disease for pre- and post-treatment core biopsies for at least 20 patients per arm on the expansion cohorts.
* Patients may have received 1-3 prior systemic therapies in the metastatic setting.
* Adequate organ function within 14 days of dosing
* Must be willing to provide and have available archival tissue for PD-L1 testing.
* Written, voluntary informed consent.
* Fertile men and women of childbearing potential must agree to use an effective method of birth control from providing signed consent and for 120 days after last study drug administration. Women of childbearing potential include pre-menopausal women and women within the first 2 years of the onset of menopause. Women of childbearing potential must have a negative pregnancy test ≤ 72 hours prior to Day 1 of study.
* Effective methods of birth control include: surgically sterile, barrier device (condom, diaphragm), contraceptive coil, intrauterine device (IUD), and abstinence.
* Life expectancy of >12 weeks.
* Patients with central nervous system disease are eligible for enrollment if they have received prior radiotherapy or surgery to sites of CNS metastatic disease and are without evidence of clinical progression for at least 4 weeks prior to screening, have no evidence of new or enlarging brain metastases, and are off steroids for at least 7 days before first dose of pembrolizumab.

Exclusion Criteria:

* Prior systemic therapy targeting PD-1: PD-L1 axis.
* Patients who are curable by conventional multidisciplinary management.
* Patients with severe and/or uncontrolled concurrent medical disease that in the opinion of the investigator could cause unacceptable safety risks or compromise compliance with the protocol.
* Patients who have received wide field radiotherapy ≤ 4 weeks or limited field radiation for palliation < 2 weeks prior to screening or who have not recovered adequately from side effects of such therapy.
* Patients who have active infections requiring therapy.
* Patients that are known to be positive for Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies), active Hepatitis B (HBsAg reactive), or Hepatitis C (HCV RNA [qualitative] is detected); patients with negative Hepatitis C antibody testing may not need RNA testing.
* Patients that have a known psychiatric or substance abuse disorder that would interfere with cooperation with the requirements of the trial.
* Patients who received systemic anti-cancer treatment prior to the first dose of study drug within the following time frames:
* Patients with active autoimmune disease or a documented history of autoimmune disease or syndrome that requires systemic steroids or immunosuppressive agents. Patients with vitiligo or resolved childhood asthma/atopy would be exception to this rule. Patients that require inhaled steroids or local steroid injections would not be excluded from the study. Patients with hypothyroidism not from autoimmune disease that is stable on hormone replacement will not be excluded from the study.
* Women who are pregnant or nursing/breastfeeding.
* Known hypersensitivity to pembrolizumab or another mAb.
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
* Patients with untreated central nervous system disease. Patients with controlled treated CNS lesions who have undergone surgery or stereotactic radiosurgery and stable for 4 weeks are eligible.
* Inability to comply with protocol required procedures.
* Patients with medical conditions that require chronic systemic corticosteroid therapy or require any other form of immunosuppressive medication. However, patients using physiologic replacement doses of hydrocortisone, or its equivalent, will be considered eligible for this study: up to 20 mg hydrocortisone (or 5 mg of prednisone) in the morning and 10 mg hydrocortisone (or 2.5 mg prednisone) in the evening.
* Patients with the risk factors for bowel obstruction or bowel perforation (examples include but not limited to a history of acute diverticulitis, intra-abdominal abscess, abdominal carcinomatosis).
* Patients who have received a live vaccine within 30 days prior to the first dose of trial treatment.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hussein Tawbi, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (12):
- United States (12):
  - University of Southern California, Los Angeles, California
  - Medstar Health Research Institute, Washington D.C., District of Columbia
  - Mayo Clinic Florida, Jacksonville, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Washington University in St. Louis, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University, Durham, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tawbi HA, Burgess M, Bolejack V, Van Tine BA, Schuetze SM, Hu J, D'Angelo S, Attia S, Riedel RF, Priebat DA, Movva S, Davis LE, Okuno SH, Reed DR, Crowley J, Butterfield LH, Salazar R, Rodriguez-Canales J, Lazar AJ, Wistuba II, Baker LH, Maki RG, Reinke D, Patel S. Pembrolizumab in advanced soft-tissue sarcoma and bone sarcoma (SARC028): a multicentre, two-cohort, single-arm, open-label, phase 2 trial. Lancet Oncol. 2017 Nov;18(11):1493-1501. doi: 10.1016/S1470-2045(17)30624-1. Epub 2017 Oct 4. PMID 28988646

RESULTS

PARTICIPANT FLOW:
Groups:
- Soft Tissue Sarcoma: Patients with the following types of soft tissue sarcoma: leiomyosarcoma, poorly differentiated/de-differentiated liposarcoma, high grade pleomorphic undifferentiated sarcoma/MFH, MPNST and synovial sarcoma). Pembrolizumab was administered at 200 mg intravenously every 3 weeks
  Pembrolizumab
- Bone Sarcoma: Patients with the following types of bone sarcoma: Ewing sarcoma, osteosarcoma, and chondrosarcoma [de-differentiated or mesenchymal]. Pembrolizumab was administered at 200 mg intravenously every 3 weeks
  Pembrolizumab
- Expansion Cohort: Patients with the following types of soft tissue sarcoma: poorly differentiated/de-differentiated liposarcoma, high grade pleomorphic undifferentiated sarcoma. Pembrolizumab was administered at 200 mg intravenously every 3 weeks
Period: Overall Study
Arm/Group | Soft Tissue Sarcoma | Bone Sarcoma | Expansion Cohort
Started | 42 | 42 | 60
Completed | 42 | 42 | 60
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Soft Tissue Sarcoma: Patients with the following types of soft tissue sarcoma: leiomyosarcoma, poorly differentiated/de-differentiated liposarcoma, high grade pleomorphic undifferentiated sarcoma/MFH, MPNST and synovial sarcoma). Pembrolizumab will be administered at 200 mg intravenously every 3 weeks
  Pembrolizumab
- Bone Sarcoma: Patients with the following types of bone sarcoma: Ewing sarcoma, osteosarcoma, and chondrosarcoma [de-differentiated or mesenchymal]. Pembrolizumab will be administered at 200 mg intravenously every 3 weeks
  Pembrolizumab
- Expansion: Patients with the following types of soft tissue sarcoma: Liposarcoma and Pleomorphic sarcoma
- Total: Total of all reporting groups
Arm/Group | Soft Tissue Sarcoma | Bone Sarcoma | Expansion | Total
Number analyzed (Participants) | 42 | 42 | 60 | 144
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 6 | 0 | 7
  Between 18 and 65 years | 32 | 34 | 38 | 104
  >=65 years | 9 | 2 | 22 | 33
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 17 | 48
  Male | 27 | 26 | 43 | 96
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 5 | 8
  Not Hispanic or Latino | 36 | 37 | 53 | 126
  Unknown or Not Reported | 4 | 4 | 2 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 2 | 1 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 2 | 4 | 9
  White | 36 | 35 | 51 | 122
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 1 | 2 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: The Objective Response Rate (ORR) is the percentage of patient's tumor that shrinks or disappears after treatment. ORR will be evaluated according to RECIST (Response Evaluation Criteria In Solid Tumors) 1.1, whereby Complete Response is defined as the disappearance of all target lesions and Partial Response is defined as at least a 30% decrease in the sum of the diameters of target lesions in reference to the baseline diameters. Overall Response (OR) = CR + PR.
Time Frame: Assessments will be conducted at 8 weeks, up to 5 years
Population: There were 40 of 42 patients in the soft tissue sarcoma cohort who were evaluable for response. There were 40 of 42 patients in the bone sarcoma cohort who were evaluable for response. There were 53 of 60 patients in the expansion cohort who were evaluable for response.
Measure: Count of Participants; unit: Participants
Arm/Group | Soft Tissue Sarcoma | Bone Sarcoma | Expansion Cohort
Number analyzed (Participants) | 40 | 40 | 53
Participants | 7 | 2 | 7
Statistical Analysis 1: Comparison: Soft Tissue Sarcoma; An objective response rate of 25% will be considered clinically meaningful and a response rate less than 10% will be considered lack of efficacy. The treatment will be considered a success if 8 or more of 40 enrolled patients have a PR or better by RECIST 1.1; Test type: Superiority — An objective response rate of 25% will be considered clinically meaningful and a response rate less than 10% will be considered lack of efficacy. The treatment will be considered a success if 8 or more of 40 enrolled patients have a PR or better by RECIST 1.1; Binomial estimate of response rate of PR = 17.5, 95% CI 2-sided [7.3 to 32.8] — Clopper-Pearson (Exact) Confidence Interval. Excluded from rate due to no response evaluation: Soft Tissue: 2; Bone: 2; Expansion: 7 patients
Statistical Analysis 2: Comparison: Bone Sarcoma; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Binomial estimate of response rate of PR = 5.0, 95% CI 2-sided [1.0 to 16.9] — Clopper-Pearson exact confidence interval; Excluded from rate due to no response evaluation: Soft Tissue: 2; Bone: 2; Expansion: 7 patients
Statistical Analysis 3: Comparison: Expansion Cohort; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Binomial estimate of response rate of PR = 13.0, 95% CI 2-sided [5.5 to 25.3] — Clopper-Pearson (Exact) Confidence Interval Excluded from rate due to no response evaluation: Soft Tissue: 2; Bone: 2; Expansion: 7 patients

2. Secondary Outcome: Adverse Events Related to Pembrolizumab Treatment in Patients With Advanced Sarcoma, by Patient
Description: Related Adverse Event is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a investigational product and related to the investigational product.
Time Frame: Up to 5 years
Measure: Number; unit: Grade 3 or higher treatment related AEs
Arm/Group | Soft Tissue Sarcoma | Bone Sarcoma | Expansion Cohort
Number analyzed (Participants) | 42 | 42 | 60
Grade 3 or higher treatment related AEs | 6 | 9 | 10

3. Secondary Outcome: The Progression-free Survival (PFS)
Description: The progression-free survival is the length of time during and after the treatment of a disease, such as cancer, that a patient lives with the disease but it does not get worse.
Time Frame: up to 5 yrs
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Soft Tissue Sarcoma | Bone Sarcoma | Expansion Cohort
Number analyzed (Participants) | 37 | 39 | 53
weeks | 18 [8 to 22] | 8 [7 to 9] | 8 [7 to 13]

4. Secondary Outcome: Response Rate by Immune-related Response Criteria (Ir-RC)
Description: Immune related response criteria was developed to adequately assess tumor response to immunotherapy.The irRC are based on bidimensional measurements We aimed to assess response by bidimensional measurements in patients with advanced sarcoma. Immune-related Complete Response (irCR) is the complete disappearance of all index lesions. Immune-related Partial Response (irPR) is the decrease by 50% or greater (from Baseline) in the sum of the products of the two largest perpendicular diameters of all index and new measurable lesions
Time Frame: Assessment at 8 weeks, up to 5 years
Population: There were 30 out of 40 total patients evaluable for response in the soft tissue sarcoma cohort. There were 30 out of 40 total patients evaluable for response in the soft tissue sarcoma cohort. There were 52 out of 60 total patients evaluable for response in the soft tissue sarcoma cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | Soft Tissue Sarcoma | Bone Sarcoma | Expansion Cohort
Number analyzed (Participants) | 30 | 30 | 52
Participants
  irCR | 1 | 0 | 2
  irPR | 2 | 2 | 7

5. Secondary Outcome: Overall Survival (OS)
Description: The Overall Survival is the length of time from either the date of diagnosis or the start of treatment for a disease, such as cancer, that patients diagnosed with the disease and are still alive
Time Frame: up to 5 years
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Soft Tissue Sarcoma | Bone Sarcoma | Expansion Cohort
Number analyzed (Participants) | 42 | 42 | 60
weeks | 49 [34 to 73] | 52 [40 to 72] | 57 [33 to 86]

ADVERSE EVENTS:
Time Frame: Adverse Event data is collected beginning from the time of treatment through 30 days following cessation of treatment or the initiation of a new anti-cancer therapy, whichever is earlier.
Groups:
- Expansion: Patients with the following types of soft tissue sarcoma: Undifferentiated pleomorphic sarcoma (UPS) and de-differentiated liposarcoma (LPS). Pembrolizumab will be administered at 200 mg intravenously every 3 weeks
Arm/Group | Soft Tissue Sarcoma | Bone Sarcoma | Expansion
All-Cause Mortality (participants affected / at risk) | 4/42 | 2/42 | 2/60
Serious Adverse Events (participants affected / at risk) | 19/42 | 15/42 | 17/60
Other Adverse Events (participants affected / at risk) | 40/42 | 42/42 | 58/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Soft Tissue Sarcoma (N=42) | Bone Sarcoma (N=42) | Expansion (N=60)
Bronchopulmonary hemmorhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Duodenal Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Neoplasms, benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 2 (2)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS - OTHER, SPECIFY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Laryngeal hemmorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nervous system disorders, other (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney inury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal and urinary disorders, other (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 2 (2) | 0 (0) | 1 (1)
Vascular disorders, other (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac disorders, other (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ventricular Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Adrenal Insufficiency (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0)
Blurred Vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colonic Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colonic Stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (1)
General Disorders and Administration site conditions (General disorders) | 0 (0) | 0 (0) | 3 (3)
Immune system disorders, other (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder, other (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Soft Tissue Sarcoma (N=42) | Bone Sarcoma (N=42) | Expansion (N=60)
Anemia (Blood and lymphatic system disorders) | 9 (9) | 8 (8) | 21 (21)
Blood and Lymphatic Systems Disorder, other (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Febrile Neuropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 2 (2)
Cardiac disorders, other (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus Tachycardia (Cardiac disorders) | 2 (2) | 2 (2) | 4 (4)
Ventricular Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ear and Labyrinth disorders, other (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Endocrine Disorders-other (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 3 (3) | 2 (2) | 2 (2)
Hypothyroidism (Endocrine disorders) | 2 (2) | 2 (2) | 7 (7)
Abdominal Pain (Gastrointestinal disorders) | 5 (5) | 1 (1) | 5 (5)
constipation (Gastrointestinal disorders) | 5 (5) | 6 (6) | 6 (6)
diarrhea (Gastrointestinal disorders) | 7 (7) | 2 (2) | 6 (6)
dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 4 (4)
flatulance (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
gastrointestinal disorders-other (Gastrointestinal disorders) | 2 (2) | 0 (0) | 4 (4)
non-cardiac chest pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
allergic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
vaginal infection (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
activated partial thromboplastin time prolonged (Investigations) | 6 (6) | 7 (7) | 8 (8)
Alanine aminotranferase increased (Investigations) | 1 (1) | 5 (5) | 4 (4)
Alkaline Phosphatase increased (Investigations) | 4 (4) | 12 (12) | 7 (7)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 7 (7) | 6 (6)
creatinine increased (Investigations) | 2 (2) | 2 (2) | 5 (5)
INR increased (Investigations) | 4 (4) | 4 (4) | 6 (6)
Lymphocyte count decreased (Investigations) | 3 (3) | 6 (6) | 10 (10)
dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 6 (6)
hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
hyperglycemia (Metabolism and nutrition disorders) | 6 (6) | 3 (3) | 8 (8)
hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (3)
hypoalbumenia (Metabolism and nutrition disorders) | 3 (3) | 5 (5) | 8 (8)
hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 4 (4)
hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 1 (1)
hyponatremia (Metabolism and nutrition disorders) | 5 (5) | 8 (8) | 8 (8)
arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 3 (3)
back pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 1 (1) | 8 (8)
chest wall pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 1 (1)
musculoskeletal and connective tissue disorder-other (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 7 (7)
pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4) | 6 (6)
tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 2 (2)
dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
headache (Nervous system disorders) | 4 (4) | 1 (1) | 2 (2)
nervous system disorders, other (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
insomnia (Psychiatric disorders) | 2 (2) | 4 (4) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
URINARY URGENCY (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 7 (7) | 7 (7)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (4) | 5 (5)
Laryngeal hemmorhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
respiratory, thoracic, and mediastinal disorders, other (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 1 (1)
erythmea multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 6 (6)
rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 7 (7)
Hot flashes (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 8 (8)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
photophobia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
gastroesophogeal reflux (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 10 (10) | 3 (3) | 9 (9)
rectal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (4) | 1 (1) | 4 (4)
chills (General disorders) | 0 (0) | 2 (2) | 5 (5)
Edema limbs (General disorders) | 3 (3) | 2 (2) | 6 (6)
Fatigue (General disorders) | 2 (2) | 1 (1) | 1 (1)
flu like symptoms (General disorders) | 0 (0) | 1 (1) | 0 (0)
general disorders-other (General disorders) | 1 (1) | 3 (3) | 5 (5)
Hypothermia (General disorders) | 0 (0) | 1 (1) | 0 (0)
localized edema (General disorders) | 0 (0) | 0 (0) | 2 (2)
malaise (General disorders) | 1 (1) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 2 (2) | 0 (0)
serum sickness (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
infections and infestations-other (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
papulopustular rash (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 4 (4)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
CPK increased (Investigations) | 0 (0) | 1 (1) | 2 (2)
investigations-other (Investigations) | 1 (1) | 3 (3) | 1 (1)
lymphocyte count increased (Investigations) | 1 (1) | 3 (3) | 1 (1)
neutrophil count decreased (Investigations) | 0 (0) | 2 (2) | 1 (1)
platelet count decreased (Investigations) | 1 (1) | 3 (3) | 3 (3)
weight loss (Investigations) | 1 (1) | 4 (4) | 0 (0)
white blood cell decreased (Investigations) | 1 (1) | 4 (4) | 0 (0)
anorexia (Metabolism and nutrition disorders) | 6 (6) | 2 (2) | 8 (8)
bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1)
joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
myalgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 2 (2)
neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
soft tissue necrosis upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
neoplasms, benign, malignant, and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
dysesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
peripheral sensory neuropathy (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1)
presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 3 (3)
depression (Psychiatric disorders) | 2 (2) | 0 (0) | 1 (1)
psychiatric disorders-other (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-09): https://cdn.clinicaltrials.gov/large-docs/39/NCT02301039/Prot_SAP_000.pdf